CLINICAL TRIAL: NCT02640105
Title: Cluster Headache (CH), Addictions and Vascular Function
Brief Title: Cluster Headache, Addictions and Vascular Function
Acronym: CHAD
Status: Completed | Type: Observational
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Other Study IDs: CHUBX 2013/14
Record Dates: First submitted 2015-11-23; First posted 2015-12-28 (Estimated); Last update posted 2022-03-31 (Actual); Status verified 2022-03

CONDITIONS: Cluster Headache
MeSH Terms: conditions — Cluster Headache | interventions — Surveys and Questionnaires; Blood Specimen Collection

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patient with Cluster headache: Prospective follow-up of patient with Cluster headache
  Interventions: Other: Neurological clinical examination; Other: Psychological clinical examination; Other: Questionnaires; Other: Blood sample; Other: Endothelial function measurement

INTERVENTIONS:
Other: Neurological clinical examination — Diagnostic and description of cluster headache
Other: Psychological clinical examination — Scale and questionnaires
Other: Questionnaires — Psychopathological and cognitive questionnaires
Other: Blood sample — Blood sample for DNA collection
Other: Endothelial function measurement — Endothelial function will be measured with a noninvasive Peripheral Arterial Tone (PAT) signal technology using the EndoPAT device

SUMMARY:
Cluster headache (CH) is one of the most painful primitive headaches. Developments in neuroimaging have demonstrated activation of the ipsilateral hypothalamic and orexinergic system, which is similar in patients with addictions. CH has strong links to the vascular system but there is no study measuring endothelial function in CH sufferers.

DETAILED DESCRIPTION:
Several studies have shown an association between Cluster headache (CH) and smoking. However, no data exists on the link between CH and other addictions, and impact of these addictions on clinical characteristics of the disease. In addition, despite the strong biological link between CH and the vascular system, systematic investigations about vascular functions in CH patients are lacking.

This will be a prospective cohort study of 150 patients with CH, conducted in the Headache Center in Bordeaux, France.

ELIGIBILITY:
Inclusion Criteria:

* Presenting a chronic or episodic cluster headache diagnosed according to the International Classification of Headache Disorders (ICH-D III) criteria, in active or inactive phase.

Exclusion Criteria:

* Other primary headaches
* Subjects without social insurance

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patient with cluster headache
Sampling Method: Non-Probability Sample
Enrollment: 95 (Actual)
Dates: Start 2014-06-25 (Actual); Primary Completion 2016-06-10 (Actual); Study Completion 2016-06-10 (Actual)

PRIMARY OUTCOMES:
Duration of active periods of cluster headache | Day 0 (Inclusion visit)
Number of active periods | Day 0 (Inclusion visit)
Duration of cluster headache | Day 0 (Inclusion visit)
Severity of attacks | Day 0 (Inclusion visit)
Duration of active periods of cluster headache | one year after inclusion
Number of active periods | one year after inclusion
Duration of cluster headache | one year after inclusion
Severity of attacks | one year after inclusion

SECONDARY OUTCOMES:
Existence of an addiction | Day 0 (Inclusion visit)
Existence of an addiction | One year after inclusion
Severity of Addiction | Day 0 (Inclusion visit)
Severity of Addiction | One year after inclusion
Reactive Hyperemic Index (RHI) | Day 0 (Inclusion visit)
  Endothelial function measurement

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France